CLINICAL TRIAL: NCT07320508
Title: A Prospective, Multicenter Study of Transarterial Epirubicin Chemotherapy in the Treatment of Sinonasal Adenoid Cystic Carcinoma
Brief Title: Epirubicin Interventional Chemotherapy for Sinonasal Adenoid Cystic Carcinoma (SNACC): A Prospective Study
Acronym: EIC-SNACC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Quan Liu, Senior doctor, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeEntFudan-2025307; 2025307 (Other: Eye and ENT Hospital, Fudan University)
Record Dates: First submitted 2025-12-12; First posted 2026-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Adenoid Cystic Carcinoma; Sinonasal Carcinoma; Epirubicin
Keywords: transarterial chemoembolization; objective response rate; 2-year progression-free surviva
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Epirubicin

STUDY DESIGN:
Intervention Model Description: This is a single-arm, response-adapted study. All enrolled participants will first receive the same interventional chemotherapy. After central imaging assessment, they will be assigned to one of two predefined, stratified local therapy pathways based on their objective tumor response (complete response or not), as per protocol.
Masking Description: This is an open-label study. The assignment to subsequent local therapy is based on objective imaging assessment (RECIST 1.1).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Chemotherapy with Epirubicin (Experimental): All participants in this single-arm study will undergo three cycles of transarterial Epirubicin chemoinfusion (60mg/m² per cycle, every 4 weeks) as the initial intervention. Following this, the imaging assessment (MRI, RECIST 1.1) will be performed. Participants will then be assigned to one of two predefined local therapy pathways based on their tumor response: those not achieving a complete response (CR) will undergo skull base surgery followed by radiotherapy; those achieving CR will receive definitive radiotherapy alone.
  Interventions: Drug: Epirubicin (E)

INTERVENTIONS:
Drug: Epirubicin (E) — Epirubicin is administered via transarterial chemoinfusion (TAI) as a neoadjuvant treatment. The drug is delivered at a dose of 60 mg/m² per cycle, diluted in normal saline at a concentration of 1 mg:1 mL. The infusion is performed through super-selective catheterization of the tumor-feeding arteries under angiographic guidance. This cycle is repeated every 4 weeks for a total of 3 cycles prior to response assessment and subsequent stratified local therapy.

SUMMARY:
This study is for patients with locally advanced sinonasal adenoid cystic carcinoma (SNACC), a rare and challenging cancer that tends to invade nerves and the skull base. The research aims to test a new precise treatment strategy. First, all participants will receive three sessions of "interventional chemotherapy" (transarterial chemoembolization) with the drug Epirubicin, which delivers high-dose chemotherapy directly to the tumor to shrink it as much as possible. About 4-6 weeks after the third session, doctors will use MRI scans to evaluate how well the tumor responded. Based on this response, patients will follow one of two personalized treatment paths: those whose tumors did not completely disappear will undergo surgery followed by radiotherapy; those whose tumors show complete disappearance on imaging will receive precise radiotherapy alone, potentially avoiding major surgery. This is a prospective, multicenter study. The main goals are to evaluate the safety and effectiveness of this response-adapted strategy and to see if it can improve outcomes for patients with this difficult-to-treat cancer.

DETAILED DESCRIPTION:
1. Background and Rationale Sinonasal adenoid cystic carcinoma (SNACC) is a rare malignancy with a propensity for perineural invasion and skull base infiltration. Complete surgical resection is challenging and often associated with significant morbidity. While systemic chemotherapy offers limited benefit, our preclinical data from patient-derived tumor organoid drug sensitivity testing identified Epirubicin as the most active agent (sensitivity rate: 87.5%, n=24).Transarterial chemoembolization allows for targeted, high-dose drug delivery to the tumor bed while minimizing systemic exposure, presenting a promising neoadjuvant strategy.
2. Study Objectives

   Primary Objectives: To evaluate the objective response rate (ORR) after three cycles of transarterial Epirubicin chemoinfusion, the 2-year progression-free survival (PFS) of the integrated strategy, and the safety profile of the interventional chemotherapy.

   Secondary Objectives: To assess the complete response (CR) rate post-chemotherapy, the safety of subsequent surgery/radiotherapy, overall survival (OS), and explore biomarkers predictive of response.
3. Study Design This is a prospective, multicenter, single-arm, interventional study. The study employs a response-adapted design.
4. Methodology

   Participants: Approximately 100 patients with histologically confirmed, locally advanced (T3/T4) SNACC will be enrolled across multiple centers in China, including [Fudan University Eye & ENT Hospital].

   Intervention: All participants will receive three cycles of transarterial Epirubicin chemoinfusion (60mg/m² per cycle, q4w). Central imaging review (MRI, RECIST 1.1) will be performed 4-6 weeks after the third cycle.

   Stratified Treatment Pathways:

   Path A (Non-CR): Patients not achieving CR will undergo planned skull base surgery followed by adjuvant radiotherapy.

   Path B (CR): Patients achieving imaging CR will proceed directly to definitive intensity-modulated radiotherapy (IMRT) without surgery.

   Assessments: Efficacy will be assessed via serial contrast-enhanced MRI. Safety will be monitored per CTCAE v5.0, including laboratory tests and cardiac function evaluation (echocardiography).

   Statistical Analysis: The sample size is calculated based on demonstrating superiority in ORR compared to a historical benchmark. PFS and OS will be analyzed using the Kaplan-Meier method. Analysis will follow the intention-to-treat principle.
5. Ethics and Dissemination The study protocol has been approved by the Institutional Review Board of [Fudan University Eye & ENT Hospital] (Approval No: [2025307]). It will be conducted in accordance with the Declaration of Helsinki. Results will be disseminated through peer-reviewed publications and academic conferences.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Histologically confirmed diagnosis of sinonasal adenoid cystic carcinoma (ACC).
3. Tumor stage T3 or T4 according to the AJCC (American Joint Committee on Cancer) 9th edition staging system. Participants with lymph node metastasis must be amenable to surgical dissection. Those with distant metastasis must have stable disease.
4. Ability to provide a sufficient volume (≥0.5 cm³) of fresh tumor tissue via biopsy or surgery for research purposes, with participant's informed consent.
5. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 to 2.
6. Voluntary participation and provision of written informed consent. Good compliance, able to cooperate with treatment and follow-up.

Exclusion Criteria:

1. Prior treatment with Epirubicin or any other anthracycline-based chemotherapy.
2. Prior radiotherapy to the head and neck region.
3. Administration of any other chemotherapy, targeted therapy, or immunotherapy within 4 weeks prior to study enrollment.
4. Concurrent participation in another interventional drug clinical trial.
5. Inadequate liver, kidney, or bone marrow function that does not meet the requirements for the planned treatment regimen.
6. Contraindications to anthracycline-containing chemotherapy regimens: known allergy to anthracyclines, presence of ≥ Grade 2 peripheral neuropathy, or uncontrolled nausea/vomiting or chronic gastrointestinal diseases.
7. Severe uncontrolled acute infection or decompensated major organ dysfunction.
8. Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-12 (Estimated); Study Completion 2029-12-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | After completion of 3 cycles (each cycle is 28 days) of interventional chemotherapy (at the time of response assessment)
  The proportion of participants achieving complete response (CR) or partial response (PR) according to RECIST 1.1 criteria, as assessed by central imaging review after completion of interventional chemotherapy.
2-year Progression-Free Survival (PFS) rate | 2 years from the start of intervention
  The proportion of participants alive without disease progression (local recurrence or distant metastasis) at 2 years from the initiation of interventional chemotherapy. Progression is defined per RECIST 1.1 criteria.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dose of interventional chemotherapy up to 30 days after the last dose (approximately 18 weeks)
  The frequency and severity of adverse events assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, specifically related to the interventional chemotherapy phase.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | After completion of 3 cycles ((each cycle is 28 days) ) of interventional chemotherapy (at the time of response assessment)
  The proportion of participants achieving complete response (CR) according to RECIST 1.1 criteria, as assessed by central imaging review after completion of interventional chemotherapy.
Incidence of Adverse Events related to Surgery and Radiotherapy | From the start of surgery or radiotherapy until 90 days after completion of local therapy
  The frequency and severity of adverse events assessed as per CTCAE v5.0, that are attributable to the subsequent local therapy (surgery and/or radiotherapy) phase of the integrated treatment.
Overall Survival (OS) | From the start of intervention, assessed up to 5 years
  The time from the initiation of interventional chemotherapy to death from any cause.
Correlation of Biomarker with Treatment Response | Tissue obtained at baseline (pre-treatment); response assessed after 3 cycles (each cycle is 28 days) of chemotherapy
  An exploratory analysis to assess the association between molecular characteristics (e.g., from tumor tissue) and objective response to Epirubicin interventional chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Liu, M.D., Principal Investigator — Eye and ENT Hospital, Fudan University
Locations (1):
- Eye and ENT Hospital, Fudan University, Shanghai, Xuhui Strict, China

IPD SHARING:
Plan to Share IPD: No
This is an investigator-initiated study conducted in China. Individual participant data (IPD) contains sensitive personal health information and is subject to strict data protection regulations in China (e.g., the Personal Information Protection Law). There is currently no approved data sharing mechanism that fully complies with these regulations while ensuring participant privacy. Therefore, there is no plan to publicly share raw IPD. Aggregate results will be shared through publication in peer-reviewed journals.

REFERENCES:
- [Result] Vermorken JB, Verweij J, de Mulder PH, Cognetti F, Clavel M, Rodenhuis S, Kirkpatrick A, Snow GB. Epirubicin in patients with advanced or recurrent adenoid cystic carcinoma of the head and neck: a phase II study of the EORTC Head and Neck Cancer Cooperative Group. Ann Oncol. 1993 Nov;4(9):785-8. doi: 10.1093/oxfordjournals.annonc.a058665. PMID 8280659
- [Result] Zhou J, Yu Z, Wang S, Li N. Practical guideline for recurrent or metastatic adenoid cystic carcinoma. Innovation (Camb). 2025 May 21;6(9):100957. doi: 10.1016/j.xinn.2025.100957. eCollection 2025 Sep 8. No abstract available. PMID 40979299
- [Result] Teymoortash A, Zieger L, Hoch S, Pagenstecher A, Hofer MJ. Distinct microscopic features of perineural invasion in adenoid cystic carcinoma of the head and neck. Histopathology. 2014 Jun;64(7):1037-9. doi: 10.1111/his.12210. Epub 2013 Aug 19. No abstract available. PMID 24033920
- [Result] van Weert S, van der Waal I, Witte BI, Leemans CR, Bloemena E. Histopathological grading of adenoid cystic carcinoma of the head and neck: analysis of currently used grading systems and proposal for a simplified grading scheme. Oral Oncol. 2015 Jan;51(1):71-6. doi: 10.1016/j.oraloncology.2014.10.007. Epub 2014 Oct 28. PMID 25456010
- [Result] Lupinetti AD, Roberts DB, Williams MD, Kupferman ME, Rosenthal DI, Demonte F, El-Naggar A, Weber RS, Hanna EY. Sinonasal adenoid cystic carcinoma: the M. D. Anderson Cancer Center experience. Cancer. 2007 Dec 15;110(12):2726-31. doi: 10.1002/cncr.23096. PMID 17960615
- [Result] Mavrikios A, Goudjil F, Beddok A, Zefkili S, Bolle S, Feuvret L, Le Tourneau C, Choussy O, Sauvaget E, Herman P, Dendale R, Calugaru V. Proton therapy and/or helical tomotherapy for locally advanced sinonasal skull base adenoid cystic carcinoma: Focus on experience of the Institut Curie and review of literature. Head Neck. 2023 Jul;45(7):1619-1631. doi: 10.1002/hed.27371. Epub 2023 Apr 25. PMID 37097003
- [Result] Bjorndal K, Krogdahl A, Therkildsen MH, Overgaard J, Johansen J, Kristensen CA, Homoe P, Sorensen CH, Andersen E, Bundgaard T, Primdahl H, Lambertsen K, Andersen LJ, Godballe C. Salivary gland carcinoma in Denmark 1990-2005: a national study of incidence, site and histology. Results of the Danish Head and Neck Cancer Group (DAHANCA). Oral Oncol. 2011 Jul;47(7):677-82. doi: 10.1016/j.oraloncology.2011.04.020. Epub 2011 May 25. PMID 21612974
- [Result] Dodd RL, Slevin NJ. Salivary gland adenoid cystic carcinoma: a review of chemotherapy and molecular therapies. Oral Oncol. 2006 Sep;42(8):759-69. doi: 10.1016/j.oraloncology.2006.01.001. Epub 2006 Jun 6. PMID 16757203

DOCUMENTS (1):
  • Study Protocol (2025-10-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT07320508/Prot_000.pdf